CLINICAL TRIAL: NCT02424682
Title: Safety of Herceptin in Metastatic Breast Cancer
Brief Title: Safety of Herceptin/Trastuzumab in Metastatic Breast Cancer
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML21201
Record Dates: First submitted 2015-04-20; First posted 2015-04-23 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Breast Cancer, Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- HER 2 positive metastatic breast cancer: HER 2 positive metastatic breast cancer treated with Herceptin as per registered indication, until disease progression.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention administered in this study

SUMMARY:
This study was designed to evaluate safety and tolerability of Herceptin as treatment for patients with human epidermal growth factor receptor 2 (HER-2) positive metastatic breast cancer. Frequency, characteristics and severity of adverse events (AE) and serious adverse events (SAE) were followed to evaluate the safety of Herceptin in patients with HER2 positive metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of metastatic breast cancer (BC) with HER2-neu overexpression
* Left Ventricular Ejection Fraction (LVEF) by ECHO or Multi Gated Acquisition Scan (MUGA) > 50%
* Good performance status: Eastern Cooperative Oncology Group (ECOG) scale < or = 2 and life expectancy > or = 12 weeks

Exclusion Criteria:

* Advanced pulmonary disease and severe dyspnea
* Abnormal laboratory within 14 days prior to registration
* Peripheral neuropathy > grade 2
* Presence of central nervous system (CNS) metastasis
* Pregnancy or lactating

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with human epidermal growth factor receptor (HER) 2 positive metastatic breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2007-08; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events (AEs) | Up to 2 years
Percentage of Participants with Serious Adverse Events (SAEs) | Up to 2 years
Percentage of Deaths | Up to 2 years

SECONDARY OUTCOMES:
Percentage of Participants with Serious Adverse Events (SAEs), Who Experienced Progression of Disease | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Kamenitz, Serbia